CLINICAL TRIAL: NCT03422211
Title: A Prospective Assessment of Opioid Utilization Post-operatively in Sports Orthopaedic Surgeries
Acronym: Opioids
Status: Completed | Type: Observational
Sponsor: St. Louis University (Other)
Responsible Party: Principal Investigator, John Capelle, MD, Medical Doctor - Researcher, St. Louis University
Other Study IDs: 28494
Record Dates: First submitted 2018-01-30; First posted 2018-02-05 (Actual); Last update posted 2021-09-24 (Actual); Status verified 2021-09

CONDITIONS: Narcotic Use; Postoperative Pain; Narcotic Abuse; Opioid Use; Opioid Abuse, Uncomplicated; Opioids; Harmful Use; Analgesic Drug Dependence; Orthopedic Disorder
MeSH Terms: conditions — Pain, Postoperative; Narcotic-Related Disorders; Opioid-Related Disorders; Musculoskeletal Diseases | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Sports orthopaedic surgery: Patients that recently underwent orthopaedic sports surgery performed by two separate surgeons
  Interventions: Other: Questionnaire

INTERVENTIONS:
Other: Questionnaire — Will ask patients questions in regards to how many narcotics they have taken and what their pain level has been.

SUMMARY:
There was a study titled "A prospective evaluation of opioid utilization after upper extremity surgical procedures: Identifying consumption patterns and determining prescribing guidelines" by Dr. Matzon and team from Thomas Jefferson University that came up with a simple set of opioid guidelines post-surgically. These guidelines are helping to guide surgeon's prescribing patterns and ideally limit the number of prescribed pain medicines. We plan to identify typical narcotic analgesic usage post sports orthopaedic surgery. We hope to identify the number of narcotic pain pills to prescribe to patients undergoing orthopaedic sports surgery in the future.

DETAILED DESCRIPTION:
1, Consent patients undergoing sports orthopaedic surgery in clinic or in pre-operative holding area and also administer first questionnaire, opioid risk tool, and pain catastrophizing scale(research) 2. Sports orthopaedic surgery (standard of care) 3. Post-op pain control regimen (standard of care) 4. Call or email patient with questionnaire every day for a week followed by weekly for 7 more weeks. The children's questionnaire will be child specific and the parent will assist the child. Will also use a picture of Wong-Baker Faces to help children identify where their pain scale is which will be given to the patient the same day that the consent is obtained to use at home(research). Questionnaire should take less than 5 minutes and will include questions about how well their pain is controlled, how many analgesic medications they have taken, and if they have tried anything else for pain. (Research) 5. Patient will continue to go to post-operative appointments as scheduled. (standard of care) 6. Will store the data from the phone calls on the secured T drive. (Research)

ELIGIBILITY:
Inclusion Criteria:

* analgesics prescribed to patient

Patients that have undergone orthopaedic sports surgeries that Dr. Kaar and Dr. Kim performed with some of the examples being:

Acromioplasty Rotator cuff repair Labral repair Proximal humerus repair versus arthroplasty Elbow instability repair Elbow arthroplasty Hip arthroscopy Hip cam lesion repair Knee arthroscopy Knee ligament repair Knee meniscus repair Achilles tendon repair Cartilage preserving procedures

Exclusion Criteria:

mental retardation inmates non-english speaking pregnant on-call trauma cases

Ages: 10 Years to 100 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Have undergone an orthopaedic sports surgery
Sampling Method: Probability Sample
Enrollment: 223 (Actual)
Dates: Start 2017-11-16 (Actual); Primary Completion 2018-11-02 (Actual); Study Completion 2018-11-02 (Actual)

PRIMARY OUTCOMES:
Number of narcotic analgesics consumed | 2 months
  Quantify narcotic analgesics

CONTACTS AND LOCATIONS:
Overall Officials: John M Capelle, MD, Principal Investigator — St. Louis University
Locations (3):
- United States (3):
  - Cardinal Glennon, St Louis, Missouri
  - Anheuser Busch Institute, St Louis, Missouri
  - SSM Health St. Mary's Hospital - St. Louis, St Louis, Missouri

IPD SHARING:
Plan to Share IPD: No
Not planning on sharing participant data in order to protect patient's confidentiality.

REFERENCES:
- [Result] Kim N, Matzon JL, Abboudi J, Jones C, Kirkpatrick W, Leinberry CF, Liss FE, Lutsky KF, Wang ML, Maltenfort M, Ilyas AM. A Prospective Evaluation of Opioid Utilization After Upper-Extremity Surgical Procedures: Identifying Consumption Patterns and Determining Prescribing Guidelines. J Bone Joint Surg Am. 2016 Oct 19;98(20):e89. doi: 10.2106/JBJS.15.00614. PMID 27869630